CLINICAL TRIAL: NCT03940950
Title: Safety and Feasibility of Intra-articular Transplantation of Autologous Adipose Derived Stromal Vascular Faction (SVF) for Treatment of Osteoarthritis of the Knee
Brief Title: Intra-articular Transplantation of Autologous Adipose Derived Stromal Vascular Faction (SVF) for Treatment of Osteoarthritis of the Knee
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Shane A. Shapiro, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-006909
Record Dates: First submitted 2019-05-06; First posted 2019-05-07 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Osteo Arthritis Knee; Degenerative Joint Disease of Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SVF (Stromal Vascular Fraction) Group (Experimental): Subjects with knee osteoarthritis (OA) will receive Autologous Adipose-Derived SVF (Stromal Vascular Fraction) cells
  Interventions: Biological: Autologous Adipose-Derived SVF (Stromal Vascular Fraction)
- Placebo Group (Placebo Comparator): Subjects with knee osteoarthritis (OA) will be treated with a placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Autologous Adipose-Derived SVF (Stromal Vascular Fraction) — 60 ml of fat is collected from subjects abdominal wall and SVF is removed from the fat. The SVF is injected into the knee through a needle.
  Arms: SVF (Stromal Vascular Fraction) Group
Drug: Placebo — Saline control that contains no active ingredient
  Arms: Placebo Group

SUMMARY:
Researchers are trying to determine the safety and feasibility of autologous, adipose derived stromal vascular fraction injections in the treatment of knee osteoarthritis

ELIGIBILITY:
Inclusion Criteria

* Male or female ages 40-75 years
* Females of childbearing potential must have a negative pregnancy test prior to receiving the study drug and will agree use adequate contraception (hormonal or barrier method or abstinence) from the time of screening to a period of 1 year following completion of the drug treatment cycle. Females of childbearing potential are defined as premenopausal and not surgically sterilized, or post-menopausal for fewer than 2 years. A urine pregnancy test will be performed prior to the administration of the study drug to confirm negative results. If the urine pregnancy test is positive, the study drug will not be administered and the result will be confirmed by a serum pregnancy test. Serum pregnancy tests will be performed at a central clinical laboratory, whereas urine pregnancy tests will be performed by qualified personnel using kit.
* Females becoming pregnant during the study will continue to be monitored for the duration of the study or completion of the pregnancy, whichever is longer. Monitoring will include perinatal and neonatal outcome. Any SAEs associated with pregnancy will be recorded. Radiographic assessment will be deferred if the patient becomes pregnant.
* Radiographic medial and/or lateral femorotibial knee OA Kellgren-Lawrence grade 2 or 3 accompanied by definite joint space narrowing as agreed upon by two study coinvestigators. If no agreement, a musculoskeletal radiologist not associated with the study will make the final grading.
* Previous 3 month or longer trial of one of the following conservative treatments: activity modification, weight loss, physical therapy, anti-inflammatory medications or injection therapy (e.g. cortisone, hyaluronic acid/viscosupplement).
* Able to routinely walk without assistance (e.g. cane, walker).
* Clinically stable target knee.
* Completed general physical evaluation with primary care provider within 12 months of enrollment.
* Fully understanding of the requirements of the study and willingness to comply with the treatment plan, including fat harvesting, laboratory tests, diagnostic imaging, repeated knee injections/aspirations, arthroscopic examination and follow-up visits and assessments.
* Can provide written informed consent and complete HIPAA documentation after the nature of the study is fully explained and prior to any study-related procedure.
* Subjects taking medications for symptomatic relief of OA under the supervision of their primary caregiver, including non-steroidal anti-inflammatory medications (e.g. COX-2 inhibitors) may continue to take these medications unless they are otherwise excluded by the protocol and as long as the dosing has been stable for 4 weeks before baseline and is anticipated to remain stable until at least 30 days following completion of the subject's treatment cycle.

Exclusion Criteria

* Pregnant or nursing, or planning on becoming pregnant during the study period.
* Congenital or acquired malformation of the target knee resulting in significant deformity or leading to problems with the study treatment or analysis of the results.
* Significant clinical malalignment requiring follow-up full length, standing X-rays.
* Orthopedic hardware or implantable devices anywhere in the body, other than dental.
* Surgery on the index knee within 1 year of study enrollment.
* Injections of any into the index knee within 3 months prior to study enrollment.
* Locking, catching, give-away or another major mechanical symptom of the target knee.
* Kellgren-Lawrence Grade 1 or-4 arthritis in the index knee.
* History of intra-articular infection in the index knee.
* History of superficial infection in the index knee within 6 months of study enrollment, or evidence of current superficial infection affecting the index knee.
* History of falls requiring medical attention, or gait instability.
* Abnormal hematology (complete blood count with differential), blood chemistry (Glucose, Calcium, Sodium, Potassium, Bicarbonate, Chloride, BUN, Creatinine, Anion Gap), or urinalysis screening laboratory results, including aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (ALP), , and CRP.. If the laboratory reports a single, non-clinically relevant, non-life-threatening result for any of these studies and is the only excluding factor it may be repeated 1 week later if the patient wishes. Normalization of that laboratory study will then be considered nonexclusionary. See Section 14.3, Appendix 3.
* Body mass index (BMI) > 40 kg/m2.
* Taking anticoagulant medications (e.g. warfarin, heparin) or clopidogrel (Plavix).
* Taking herbal therapies or supplements within 4 weeks of enrollment or unwilling to avoid use of herbal therapies or supplements until at least 30 days following completion of the study drug treatment cycle (includes, but not limited to chondroitin sulfate, diacerein, n-glucosamine, piascledine, and capsaicin).
* Taking non-steroidal anti-inflammatory medications (e.g. COX-2 inhibitors) without a stable dosing regimen for at least 4 weeks before baseline evaluation, or anticipating not remaining on a stable dose until at least 30 days following completion of the study drug treatment cycle.
* Use of electrotherapy or acupuncture for OA, unless there is a stable regimen for at least 4 weeks before baseline assessment.
* Taking anti-rheumatic disease medication (including methotrexate or other antimetabolites) within 3 months prior to study enrollment.
* On chronic, immunosuppressive transplant therapy or having a chronic, immunosuppressive state, including use of systemic steroids/corticosteroids.
* Current tobacco product use, including nicotine patch or other nicotine products.
* Systemic inflammatory, rheumatological or connective tissue disorder including but not limited to rheumatoid arthritis, systemic sclerosis, system lupus erythematosus, and Ehlers-Danlos Syndrome.
* Rheumatological or inflammatory disease of the knee or chondrocalcinosis/calcium pyrophosphate disease (CPPD), hemochromatosis, inflammatory arthritis, arthropathy of the knee associated with juxta-articular Paget's disease of the femur or tibia, ochronosis, hemophilic arthropathy, infectious arthritis, Charcot's knee joint, villonodular synovitis, and synovial chondromatosis.
* Ongoing infectious disease, including but not limited to tuberculosis, HIV, hepatitis, and syphilis.
* Clinically significant cardiovascular (e.g. history of myocardial infarction, congestive heart failure or uncontrolled hypertension > 90 mmHg diastolic and/or 180 mmHg systolic), neurologic (e.g. stroke, TIA) renal, hepatic, orthopedic (e.g. surgery on other weight bearing joints that will interfere with study, osteoporosis, acute lower body fractures), or endocrine disease (e.g. diabetes).
* Vascular or neurological disorder affecting the index either lower limb.
* History of cancer/malignancy with the exception of adequately treated basal cell or squamous cell carcinoma of the skin not associated with the target knee within the last 5 years.
* History of blood dyscrasia, including but not limited to anemia, thrombocytopenia, and monoclonal gammopathy.
* Participation in a study of an experimental drug or medical device within 3 months of study enrollment.
* Known allergy to local anesthetics of other components of the study drug.
* Any contraindication to MRI scan according to MRI guidelines, or unwillingness to undergo MRI procedures.
* History of or current evidence of alcohol or drug abuse or dependence, recreational use of illicit drug or prescription medications, or have use of medical marijuana within 30 days of study entry.
* Any illness or condition which, in the investigators' judgement will interfere with the patient's ability to comply with the protocol, compromise patient safety, or interfere with the interpretation of the study results.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-07-02 (Actual); Primary Completion 2025-05-05 (Actual); Study Completion 2025-05-23 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 2 years
  Number of adverse events reported

CONTACTS AND LOCATIONS:
Overall Officials: Shane A Shapiro, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials